CLINICAL TRIAL: NCT00220740
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Efficacy and Safety of IGIV-Chromatography (IGIV-C), 10% Treatment in Subjects With Chronic Inflammatory Demyelinating Polyneuropathy
Brief Title: Immune Globulin Intravenous (IGIV) For Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Acronym: ICE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100538
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
Keywords: Immunoglobulin G
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — gamma-Globulins; Caprylates; Immunoglobulins, Intravenous; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): IGIV-C
  Interventions: Drug: Immune Globulin IV (Human), 10% Caprylate/Chromatography Purified
- Group 2 (Placebo Comparator)
  Interventions: Drug: Albumin (Human) 25%, United States Pharmacopeia (USP)

INTERVENTIONS:
Drug: Immune Globulin IV (Human), 10% Caprylate/Chromatography Purified — 2 g/kg body weight ideally over 2-4 days . Thereafter, study drug infusion (IGIV-C) will be administered every 3 weeks at a dose of 1 g/kg bw, given over 1-2 days for a total of 7 additional infusions
  Other Names: IGIV-C; IGIV-Chromatography (IGIV-C), 10%; Gamunex®; Gaminex®; IGIVnex; Intravenous Immunoglobulin (Human) (IGIV); Intravenous Immunoglobulin (Human); IVIG; IGIV; Intravenous Immune Globulin (Human); TAL-05-00004; Bay 41-1000; NDC13533-645-12; NDC13533-645-15; NDC13533-645-20; NDC13533-645-71; NDC13533-645-24
  Arms: Group 1
Drug: Albumin (Human) 25%, United States Pharmacopeia (USP) — Albumin 25%, USP diluted with dextrose 5% to a final concentration of 0.1% as an intravenous infusion. Alternatively, it may be a bottled placebo of 0.1% Albumin (Human) in 0.2 M Glycine, 1.1 mm sodium caprylate, 0.25% sodium chloride. 2 g/kg body weight ideally over 2-4 days . Thereafter, infusion (placebo) will be administered every 3 weeks at a dose of 1 g/kg bw, given over 1-2 days for a total of 7 additional infusions
  Other Names: Albumin (Human) 25%, USP; Plasbumin®-25; Plasbumin®-25 (Low Aluminum); TAL-05-00009; TAL-05-00025; Bay 34-9255; NDC 13533-684-16; NDC 13533-684-20; NDC 13533-684-71; NDC 13533-692-16; NDC 13533-692-20; NDC 13533-692-71
  Arms: Group 2

SUMMARY:
The intent of this study is to demonstrate the efficacy and safety of Immune Globulin Intravenous (Human), 10% Caprylate/Chromatography Purified (IGIV-C) in newly or previously diagnosed CIDP subjects. Eight courses of treatment with either placebo or IGIV-C will occur every 3 weeks. Neurological function will be measured by Inflammatory Neuropathy Cause and Treatment (INCAT) scores. Patients who deteriorate or show no improvement between day 16 and month 6 will receive the alternate study drug for an additional 6 months.

DETAILED DESCRIPTION:
110 subjects, 55 per treatment group, with newly or previously diagnosed CIDP defined by INCAT neurophysiological diagnostic criteria will be enrolled into the trial. Patients will not be replaced if they discontinue prematurely.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CIDP must be made by a neurologist specializing/experienced in neuromuscular diseases based on: a) Progressive or relapsing motor and sensory dysfunction of more than one limb resulting from neuropathy over the 2 months prior to the date informed consent is obtained, and b) Cerebrospinal fluid (CSF) less than 50 white cells/µl since CIDP diagnosis (CSF testing studies are NOT mandatory)
* Fulfillment of INCAT neurophysiological criteria for focal demyelinating polyradiculoneuropathy
* Overall INCAT score between 2-9 and significant disability in upper or lower limb function in at least 2 limbs. (An INCAT score of 2 must be exclusively from leg disability to qualify.)

Exclusion Criteria:

* Treatment with IGIV or plasma within 3 months prior to entry
* Steroids (Prednisolone or equivalent) > 10 mg/day or equivalent (i.e., > 20 mg every 2 days) during the last 3 months prior to entry
* Treatment with immunomodulatory/immunosuppressive agents (azathioprin, tacrolimus,cyclosporin, Muromonab-CD3 (OKT3), any interferon), previous lymphoid irradiation or prior treatment with cyclophosphamide, methotrexate, mitoxantrone or any other immunosuppressant drug within the past 6 months prior to entry
* Concomitant use of supplements containing any amount of fish oil within 30 days prior to entry
* Respiratory impairment requiring mechanical ventilation
* Myelopathy or evidence of central demyelination or persisting neurological deficits from stroke, central nervous system (CNS) trauma or peripheral neuropathies of other cause which include diabetes mellitus (defined as a history of type 1 or type 2 diabetes with fasting plasma glucose ≥ 7.0 mmol/L), uremic, toxic and familial neuropathies
* Pure motor syndrome fulfilling criteria for multifocal motor neuropathy with conduction block. Lower motor neuron disorder with motor weakness in an upper limb, without sensory deficit and with proximal conduction block (50% decrease in amplitude/area with proximal distal stimulation ) in motor nerves and normal sensory nerve conduction studies.
* Clinical or known evidence of associated systemic diseases that might cause neuropathy, including but not limited to connective tissue disease, HIV infection, hepatitis, Lyme disease, cancer (with the exception of benign skin cancer), Castleman's disease and systemic lupus erythematosus, diabetes mellitus (defined as a history of type 1 or type 2 diabetes with fasting plasma glucose ≥ 7.0 mmol/L), a malignant plasma cell dysplasia, immunoglobulin M (IgM) paraproteinemia, and amiodarone therapy.
* History of anaphylaxis or severe systemic response to immunoglobulin or with a blood product.
* Cardiac insufficiency (NYHA III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease, or history of congestive heart failure, severe hypertension (diastolic pressure >120 mmHg or systolic >170 mmHg).
* Females who are pregnant, breast feeding, or if of childbearing potential, unwilling to practice adequate contraception throughout the study.
* Known hyperviscosity.
* History of renal insufficiency or serum creatinine levels > 221 µmol/L (2.5 mg/dL).
* Known selective immunoglobulin A (IgA) deficiency.
* Other investigational drugs received within the 30 days prior to entry
* Conditions whose symptoms and effects could alter protein catabolism and/or immunoglobulin G (IgG) utilization (e.g. protein-losing enteropathies, nephrotic syndrome).
* Known hypercoagulable state.
* Mentally challenged adult subjects who cannot give independent informed consent.
* Subjects with uncompensated hypothyroidism (abnormally high thyroid-stimulating hormone (TSH) and abnormally low T4) or vitamin B12 deficiency (abnormally low) within the last 3 months prior to entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2004-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Latov, MD, Principal Investigator — Columbia University
Locations (32):
- United States (6):
  - Yale University School of Medicine, New Haven, Connecticut
  - Saint Louis University Medical Center, St Louis, Missouri
  - Columbia University, New York, New York
  - Wake Forest University-School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas-Southwestern Medical Center at Dallas, Dallas, Texas
- Argentina (4):
  - Hospital Ramos Mejia, Buenos Aires
  - Hospital Frances, Buenos Aires
  - Fundacion para la Lucha contra Las Enfermedades Neurologicas de la Infacia (FLENI), Buenos Aires
  - Instituto de Neurociencias Buenos Aires (INEBA), Capital Federal
- Vancouver Hospital and Health Sciences Center, Vancouver, British Columbia, Canada
- Czechia (4):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice Ostrava, Ostrava-Poruba
  - Neurologická klinika Pardubice, Pardubice
  - Fakultní nemocnice Motol, Prague
- Jüdisches Krankenhaus, Berlin, Germany
- Israel (3):
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofe Medical Center, Zrifin
- Italy (3):
  - Dipartimento di Neuroscienze, Sezione di Neurologia, AO Chieti, Chieti
  - Univesita delgi Studi di Genova, Dipartimento di Scienze, Neurologiche e della Visione, Genova
  - Hospital San Raffaele, Milan
- Mexico (3):
  - Antiguo Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Hospital Angel Leano, Neurology Department, Guadalajara, Jalisco
  - Hospital Central San Luis Potosi, Neurology Department, San Luis Potosí City
- Poland (6):
  - County Specialist Hospital, Neurology Department, Gdansk
  - Centre of Clinical Neurology, Neurology Department, Krakow
  - Barlicki Hospital, Lodz
  - Medical Acedemy, Clinical Hospital, Neurology Department, Lubin
  - Central Clinical Hospital, Medical Academy Warsaw, Warsaw
  - County Hospital, Zgierz
- University Hospital, University of Belgrade, Belgrade, Serbia

REFERENCES:
- [Result] Hughes RA, Donofrio P, Bril V, Dalakas MC, Deng C, Hanna K, Hartung HP, Latov N, Merkies IS, van Doorn PA; ICE Study Group. Intravenous immune globulin (10% caprylate-chromatography purified) for the treatment of chronic inflammatory demyelinating polyradiculoneuropathy (ICE study): a randomised placebo-controlled trial. Lancet Neurol. 2008 Feb;7(2):136-44. doi: 10.1016/S1474-4422(07)70329-0. PMID 18178525
- [Result] Bril V, Katzberg H, Donofrio P, Banach M, Dalakas MC, Deng C, Hanna K, Hartung HP, Hughes RA, Latov N, Merkies IS, van Doorn PA; ICE Study Group. Electrophysiology in chronic inflammatory demyelinating polyneuropathy with IGIV. Muscle Nerve. 2009 Apr;39(4):448-55. doi: 10.1002/mus.21236. PMID 19260050
- [Result] Merkies IS, Bril V, Dalakas MC, Deng C, Donofrio P, Hanna K, Hartung HP, Hughes RA, Latov N, van Doorn PA; ICE Study Group. Health-related quality-of-life improvements in CIDP with immune globulin IV 10%: the ICE Study. Neurology. 2009 Apr 14;72(15):1337-44. doi: 10.1212/WNL.0b013e3181a0fd80. PMID 19365055
- [Result] Hughes RA. Intravenous immunoglobulin for chronic inflammatory demyelinating polyradiculoneuropathy: the ICE trial. Expert Rev Neurother. 2009 Jun;9(6):789-95. doi: 10.1586/ern.09.30. PMID 19496683
- [Derived] Donofrio PD, Bril V, Dalakas MC, Deng C, Hanna K, Hartung HP, Hughes R, Latov N, Merkies I, van Doorn P; IGIV-C CIDP Efficacy (ICE) Study Group. Safety and tolerability of immune globulin intravenous in chronic inflammatory demyelinating polyradiculoneuropathy. Arch Neurol. 2010 Sep;67(9):1082-8. doi: 10.1001/archneurol.2010.223. PMID 20837852
- [Derived] Merkies IS, van Nes SI, Hanna K, Hughes RA, Deng C. Confirming the efficacy of intravenous immunoglobulin in CIDP through minimum clinically important differences: shifting from statistical significance to clinical relevance. J Neurol Neurosurg Psychiatry. 2010 Nov;81(11):1194-9. doi: 10.1136/jnnp.2009.194324. Epub 2010 Jul 20. PMID 20647554
- [Derived] Latov N, Deng C, Dalakas MC, Bril V, Donofrio P, Hanna K, Hartung HP, Hughes RA, Merkies IS, van Doorn PA; IGIV-C CIDP Efficacy (ICE) Study Group. Timing and course of clinical response to intravenous immunoglobulin in chronic inflammatory demyelinating polyradiculoneuropathy. Arch Neurol. 2010 Jul;67(7):802-7. doi: 10.1001/archneurol.2010.105. Epub 2010 May 10. PMID 20457948
- See also: FDA Approved Product Labeling Information - Gamunex® — http://www.talecris-pi.info/inserts/gamunex.pdf
- See also: FDA Approved Product Labeling Information - Plasbumin®-25 (Low Aluminum) — http://www.talecris-pi.info/inserts/plasbumin25la.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 study centers in USA, Poland, Argentina, Czech Republic, Canada, Mexico, Italy, Israel, Germany, and Serbia.
Groups:
- IGIV-C: 2 g/kg loading dose, followed by 1 g/kg maintenance dose
- Placebo: .1% albumin; 2g/kg loading dose and 1 g/kg maintenance dose
Period: Efficacy Period
Arm/Group | IGIV-C | Placebo
Started | 59 | 58
Completed | 33 | 12
Not Completed | 26 | 46
Not completed — Entered rescue treatment with placebo | 23 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Entered Rescue Treatment with IGIV-C | 0 | 45
Period: Rescue Treatment
Arm/Group | IGIV-C | Placebo
Started | 45 (Only the subjects who failed the treatment in the Efficacy period entered the Rescue period.) | 23 (Only the subjects who failed the treatment in the Efficacy period entered the Rescue period.)
Completed | 26 | 5
Not Completed | 19 | 18
Period: Withdrawal Period
Arm/Group | IGIV-C | Placebo
Started | 43 (The subjects who were success in Efficacy or Rescue Period were re-randomized to Withdrawal period.) | 31 (The subjects who were success in Efficacy or Rescue Period were re-randomized to Withdrawal period.)
Completed | 37 | 16
Not Completed | 6 | 15

BASELINE CHARACTERISTICS:
Groups:
- Placebo: .1% albumin, 2 g/kg loading dose, followed by 1 g/kg maintenance dose
- Total: Total of all reporting groups
Arm/Group | IGIV-C | Placebo | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 44 | 40 | 84
  >=65 years | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (17.31) | 53.3 (15.63) | 51.6 (16.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 12 | 40
  Male | 31 | 46 | 77
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6
  Czech Republic | 7 | 6 | 13
  Mexico | 3 | 5 | 8
  Canada | 1 | 1 | 2
  Argentina | 8 | 7 | 15
  Poland | 15 | 15 | 30
  Israel | 8 | 7 | 15
  Germany | 2 | 3 | 5
  Italy | 6 | 6 | 12
  Macedonia, The Former Yugoslav Republic of | 5 | 6 | 11
Baseline INCAT Score [Mean (Standard Deviation); unit: units on a scale] — Baseline INCAT score for all subjects and subgroups for Efficacy Period, Rescue treatment, and Randomized Withdrawal Period (ITT population) Measurements are reported in Inflammatory Neuropathy Case And Treatment (INCAT) scale of 0-5 in both lower and upper extremities, for a total score of 0 to 10.
  INCAT scores for arm disability: 0 = no upper limb problems; 5 = inability to use either arm for any purposeful movement.
  INCAT scores for leg disability: 0= walking not affected; 5 = restricted to wheelchair, unable to stand and walk a few steps with help
  units on a scale
    Total Overall Disability Score | 4.2 (1.4) | 4.1 (1.5) | 4.2 (1.4)
    Upper Extremity Disability Score | 2.3 (1.0) | 2.1 (1.0) | 2.2 (1.0)
    Lower Extremity Disability Score | 1.9 (0.8) | 1.9 (1.1) | 1.9 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Responder Rates Between Two Treatment Groups in the Efficacy Period
Description: The primary efficacy objective was the comparison of IGIV-C and Placebo group Responder rates. An Efficacy Period Responder was defined as a subject with ≥ 1 point improvement in the adjusted Inflammatory Neuropathy Case And Treatment (INCAT) score, with the improvement maintained through the end of Week 24 in the Efficacy Period.
  Measurements are reported in INCAT scale of 0-5 in both lower and upper extremities, for a total score of 0 to 10.
  INCAT scores for arm disability: 0 = no upper limb problems; 5 = inability to use either arm for any purposeful movement.
  INCAT scores for leg disability: 0= walking not affected; 5 = restricted to wheelchair, unable to stand and walk a few steps with help
Time Frame: 6 months
Population: The Intent-to-Treat Population was defined as all randomized subjects. This population was the primary efficacy population to be analyzed.
Measure: Number; unit: percentage of responders
Arm/Group | IGIV-C | Placebo
Number analyzed (Participants) | 59 | 58
percentage of responders | 54.2 | 20.7
Statistical Analysis 1: Comparison: IGIV-C vs Placebo; The primary efficacy endpoint was the comparison of the Responder rates in the ITT population. Treatment group differences were tested by a Chi-square test. Subjects who did not complete the 24 week Efficacy Period and entered Rescue treatment with the alternative treatment were counted as Nonresponders; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Mean Change in the Amplitude (Millivolts) in the Most Severely Affected Motor Nerve During the Efficacy Period
Description: Mean changes in amplitude [mV] measured at most proximal site in the most severely affected motor nerve from baseline to endpoint during the Efficacy Period (Intent to treat population)
Time Frame: 6 months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Millivolts
Arm/Group | IGIV-C | Placebo
Number analyzed (Participants) | 59 | 58
Millivolts | 0.69 (1.856) | 0.47 (2.291)
Statistical Analysis 1: Comparison: IGIV-C vs Placebo; Test type: Superiority or Other; p = 0.542, ANCOVA

3. Secondary Outcome: Mean Change in Grip Strength During the Efficacy Period
Time Frame: 6 months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: kilopascal
Arm/Group | IGIV-C | Placebo
Number analyzed (Participants) | 59 | 58
kilopascal
  Dominant hand (IGIV-C n=57, Placebo n=58) | 13.175 (19.2935) | 1.489 (15.5742)
  Non-dominant hand (IGIV-C n=58, Placebo n=58) | 13.316 (17.3526) | 4.261 (14.8959)
Statistical Analysis 1: Comparison: IGIV-C vs Placebo; Dominant hand; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: IGIV-C vs Placebo; Non-dominant hand; Test type: Superiority or Other; p = 0.005, ANCOVA

4. Secondary Outcome: Time to Relapse for Subjects Who Were IGIV-C Responders or IGIV-C Rescue Successes, During the Randomized Withdrawal Period
Time Frame: 6 months
Population: In the Randomized Withdrawal Period, 43 subjects were randomized to IGIV-C, but only 31 out of the 41 subjects were prior IGIV-C responders or rescue successes. Similarly, 31 subjects were randomized to Placebo, but only 26 out of the 31 subjects were prior IGIV-C responders or rescue successes.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | IGIV-C | Placebo
Number analyzed (Participants) | 31 | 26
weeks | 21.89 (6.181) | 16.56 (8.543)

ADVERSE EVENTS:
Groups:
- IGIV-C: 2 g/kg loading dose, followed by 1 g/kg maintenance dose.
  A total of 113 subjects were exposed to IGIV-C across all three treatments/periods.
- Placebo: .1% albumin; 2g/kg loading dose and 1 g/kg maintenance dose.
  A total of 95 subjects were exposed to Placebo across all three treatments/periods.
Arm/Group | IGIV-C | Placebo
Serious Adverse Events (participants affected / at risk) | 6/113 | 8/95
Other Adverse Events (participants affected / at risk) | 81/113 | 25/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C (N=113) | Placebo (N=95)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Medical observation (for asthma) (Investigations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
CIDP (relapse) (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C (N=113) | Placebo (N=95)
Nausea (Gastrointestinal disorders) | 7 (9) | 3 (3)
Pyrexia (General disorders) | 14 (26) | 0 (0)
Asthenia (General disorders) | 9 (10) | 3 (4)
Chills (General disorders) | 9 (10) | 0 (0)
Influenza (Infections and infestations) | 6 (6) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 1 (1)
Headache (Nervous system disorders) | 34 (55) | 8 (15)
Dizziness (Nervous system disorders) | 6 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 8 (13) | 1 (1)
Hypertension (Vascular disorders) | 10 (20) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must send a draft manuscript of the publication or abstract to the sponsor thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion between the sponsor and the investigator(s), the contents of the publication will be discussed in order to find a solution that satisfies both parties.